CLINICAL TRIAL: NCT01230606
Title: Ambulatory Closure Device Percutaneous Intervention: a Multi-Center Randomized Trial Evaluating Patient Satisfaction, Safety, and Cost Effectiveness of Ambulatory PCI in the Current Era
Brief Title: Same Day Versus Next Day Discharge: Ambulatory Closure Device Percutaneous Intervention
Acronym: ABCD-PCI
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Dr. Michael C. Kim, Mount Sinai School of Medicine
Other Study IDs: GCO 07-1324
Record Dates: First submitted 2010-03-31; First posted 2010-10-29 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Cardiovascular Disease
Keywords: Percutaneous Intervention; Percutaneous Coronary Intervention; Catheterization; Coronary Catheterization; Same day Discharge; Next Day Discharge; Patient Satisfaction; Multi-Center; Randomized; Low-risk PCI; BlindedClosure device; Vascular closure device
MeSH Terms: conditions — Cardiovascular Diseases; Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- overnight: Subjects that stay overnight at the hospital.
  Interventions: Other: discharge vs. overnight stay
- Next Day Discharge: Subjects that are discharged on the same day of the procedure.
  Interventions: Other: discharge vs. overnight stay

INTERVENTIONS:
Other: discharge vs. overnight stay — At six hours post-PCI,patients will be randomized to be discharged immediately or to stay overnight in the hospital for observation and discharged the following day. Randomization will occur in a 1:1 ratio. Additionally, randomization will be performed stratified by study site.

SUMMARY:
This is a multi-center trial that will evaluate the safety, feasibility, and cost effectiveness of discharging patients, who have had successful percutaneous coronary intervention (PCI) and deployment of the AngiomaxTM closure device, 6 hours after against 24 hours after the procedure. Patients will be randomized in a 3 (test): 1 (control) fashion and will have a study population of 600 patients over 6 investigational sites all within the United States. Patients <65 years old will be chosen in order to stay within the low risk group and will be followed up after 24 hours, 7 days, and 30 days via phone or office visit. The primary endpoint will be a composite of major adverse cardiac and cerebral events, and the incidence of major bleeding or vascular complications. Data acquired from the study, such as blinded financial information and patient satisfaction surveys, will be used in order to evaluate cost analysis and safety of the procedure.

DETAILED DESCRIPTION:
Closure devices are a relatively new method for sealing the femoral arterial puncture following procedures including percutaneous intervention (PCI). Because the risk of severe complications (e.g., bleeding, myocardial infarction, stroke, and mortality) associated with PCI when closure devices are very low, many patients undergoing PCI may be considered eligible for a same day hospital discharge. As the practice of ambulatory PCI is becoming more common, it is important to evaluate the readiness of patients under-going PCI for same-day discharge and anxiety and coping abilities of patients post-discharge. Our hypothesis is that same day discharge of patients who have undergone a PCI procedure with closure using a vascular closure device is safe, patients will be comfortable with a same day discharge and this process will be more cost efficient than the current standard of staying in the hospital overnight. The current pilot study is a multi-center, randomized parallel arm, controlled trial of low-risk patients undergoing an elective PCI procedure. Overall, 600 patients will be enrolled. After providing informed consent, participants will be randomized to leave the hospital on the same day as the PCI procedure or stay overnight in a 1:1 ratio. Data collection includes a self-administered questionnaire at hospital discharge, telephone interviews at 7-days and 30-days post-hospital discharge, and chart abstraction. The primary outcome for this study is differences across randomization arm in patient satisfaction scores on the validated 10-item Post-discharge coping difficulty scale assessed 7 days post-discharge. Secondary outcomes will include differences across randomization group for symptoms of anxiety, readiness for hospital discharge, patient satisfaction with the timing of their discharge, post-procedure pain and soreness, and cost-savings. While a data safety monitoring board will track all adverse events (i.e., myocardial infarction, hematoma, hospitalizations, and mortality), we anticipate too few events to occur to make meaningful inferences beyond that PCI is safe regardless of the timing of hospital discharge. The data from this pilot study will determine the comfort patients experience after undergoing PCI with an ambulatory (i.e, same-day) hospital discharge. Furthermore, this pilot study will provide the foundation for a large scale non-inferiority study of same-day discharge on outcomes including myocardial infarction, bleeding, and mortality. Such data will indicate the overall feasibility of early ambulatory PCI and has the potential to radically alter health care delivery following PCI.

ELIGIBILITY:
Inclusion Criteria:

. <75 years of age at the time of procedure.

2. Patient has a type A or B lesion(s)

3. Femoral access site is amenable to closure with a vascular closure device.

4. Over 2 hours since the completion of the PCI procedure (at least 2 hours must elapse from completion of the PCI before subjects become eligible).

Exclusion Criteria:

1. Patient has a life expectancy less than 12 months.
2. Patient has recent evidence of an acute coronary syndrome (MI)
3. Femoral access is difficult or site is not amenable to closure device
4. Anticoagulants other than unfractionated heparin or bivalirudin were used during the procedure (i.e. enoxaparin).
5. Patient has sub optimal angiographic outcome or clinical complication(s) during PCI
6. The PCI occurred in something other than a native coronary artery
7. Angiographic evidence of thrombus
8. Patient has more than 3 stents implanted during this PCI
9. Patient has an INR >2, Platelet count <100,000 or Hematocrit <25
10. Occlusion of major side branch during PCI of >1.5mm
11. Patient has ejection fraction ≤30%
12. Known allergy to PCI procedural medications
13. Patient reports living further than 30 minutes from a hospital by ambulance.
14. Patient provides informed consent and agrees to the follow-up schedule.
15. Evidence of vascular complication(s) (e.g. dissection, hematoma, bleeding) peri-procedure
16. Patient is pregnant
17. Evidence of infection (e.g. fever, pus, swelling) peri-procedure
18. Patients with chronic renal insufficiency (e.g. serum creatinine ≥1.5 mg/dL)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study will include patients undergoing an elective PCI. Overall, 600 patient will be recurited from two sites in the United Sates. As this is a feasiblity study, enrollment will be restricted to low-risk patients. For this reason, the study will be limited to patients under 75 years of age. All patients must meet all of the inclusion criteria and have none of the exclusion criteria to be enrolled into the study.
Sampling Method: Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Post-hospitalization patient satisfaction | 30 days after enrollment
  The primary endpoint is the difference in post-hospitalization patient satisfaction during the initial seven days following PCI. Post-hospitalization patient satisfaction will be assessed using the 10-item Post-Discharge Coping Difficulty scale.

SECONDARY OUTCOMES:
Patient satisfaction with timing of discharge | 30 days after enrollment
  Secondary outcomes will include post-hospital anxiety, readiness for hospital discharge, patient satisfaction with the timing of their discharge, post-procedure pain and soreness, resource utilization and cost-savings.
Patient Satisfaction Outcome Assessment | 30 days After Enrollment
  These outcomes will be assessed using standardized questionnaires and validated techniques. The composite of major adverse cardiac events (MACE) and cerebral events and the incidence of major bleeding or vascular complications will be monitored for all patients through the 30 day follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Kim, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai School of Medicine, New York, New York
  - Baylor University Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Kim M, Muntner P, Sharma S, Choi JW, Stoler RC, Woodward M, Mann DM, Farkouh ME. Assessing patient-reported outcomes and preferences for same-day discharge after percutaneous coronary intervention: results from a pilot randomized, controlled trial. Circ Cardiovasc Qual Outcomes. 2013 Mar 1;6(2):186-92. doi: 10.1161/CIRCOUTCOMES.111.000069. Epub 2013 Mar 12. PMID 23481528